CLINICAL TRIAL: NCT06488950
Title: A Study Study of Tumor Infiltrating Lymphocytes Injection (GC101/203 TIL) in Patients With Advanced Solid Tumors
Brief Title: A Study of TIL in Advanced Solid Tumors (DFGD)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC101/203-2023-DFGD-ST
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor; Tumor Infiltrating Lymphocytes; Treatment Side Effects; Effects of Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm B (Experimental): GC203 TILs will be infused i.v. to patients with advanced solid tumors after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: GC203 TIL(gene-edited TIL) or autologous TILs
- Arm A (Experimental): GC101 TILs will be infused i.v. to patients with advanced solid tumors after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: GC203 TIL(gene-edited TIL) or autologous TILs

INTERVENTIONS:
Biological: GC203 TIL(gene-edited TIL) or autologous TILs — the candidates will be assigned to GC203 TIL(gene-edited TIL) group or autologous TILs group according the volume of TIL sample

SUMMARY:
This study is to investigate the safety and efficacy of tumor infiltrating lymphocyte (TIL) therapy in patients with advanced solid tumors. Autologous TILs and gene-edited TILs are expanded from tumor resections or biopsies and infused i.v. into the patient after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* have one the tumor resection for TILs production and successfully produced；
* Age: 18 years to 75years;
* Histologically diagnosed as solid tumors;
* Expected life-span more than 3 months;
* ECOG score 0-1;
* Test subjects have failed standard treatment regimens, and be willing to receive TIL therapy;
* At least 1 evaluable tumor lesion;

Exclusion Criteria:

* with other malignant tumors, except for the malignancies that have been cured, have been inactive for ≥5 years prior to study inclusion and have a very low risk of recurrence; Non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence; Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
* Need glucocorticoid treatment, and daily dose of Prednisone greater than 10mg(or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
* Breathe indoor air in a quiet state, and the oxygen saturation of finger pulse is < 95%;
* Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
* Significant cardiovascular anomalies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  To characterize the safety profile of TILs in patients with advanced solid tumors who were failed to standard treatment as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease Control Rate (DCR） | Up to 36 months
  Percentage of patients that meet CR, PR and SD criteria set in this study according to RECIST 1.1
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time length between TIL infusion and confirmed subsequent disease progression according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Qian Zhang, Principal Investigator — Eastern Hepatobiliary Surgery Hospital; Wenlong Yu, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Third Affiliated Hospital of Naval Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes